CLINICAL TRIAL: NCT06469970
Title: INDICIA: Evolution of the Initial Distribution Volume of Glucose in the Severe Burned Adults
Brief Title: Evolution of the Initial Distribution Volume of Glucose in the Severe Burned Adults
Acronym: INDICIA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-03-CHRMT
Record Dates: First submitted 2024-06-14; First posted 2024-06-24 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2024-12

CONDITIONS: Burns; Intensive Care; Emergencies
MeSH Terms: conditions — Burns; Emergencies | interventions — Glucose

STUDY DESIGN:
Intervention Model Description: This is a prospective, observational, single-centre phase II (exploratory) cohort study aiming to describe changes in initial distribution volume of glucose (IDVG) during the first 4 days of care for patients with severe burns. Patients will be included on admission to the Burn Treatment Centre and IDVG will be measured on admission, then every 8 hours for the first 24 hours of the stay, then every 24 hours until the fourth day. The rest of the evaluation criteria correspond to standard practice in the management of severely burned patients according to the department's procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glucose administration (Experimental)
  Interventions: Drug: Glucose 30% Intravenous Solution

INTERVENTIONS:
Drug: Glucose 30% Intravenous Solution — Measurement of IDVG on admission, at 4 hours (H+4), and at 8, 16, 24, 48, 72 and 96 hours (H+8, H+16, H+24, H+48, H+72 and H+96) post-burn. The principle of this measurement consists of taking a reference blood glucose level measured on an arterial blood sample (arterial catheter) using a blood glucose meter. A bolus of 5g of glucose is injected into a central venous line over 30 seconds. A second blood glucose level is measured 3 minutes after the end of the injection.
  The intra-thoracic blood volume (ITBV) and extra-vascular lung water (EVLW) are measured using the PiCCO device as part of the usual management of burn patients.

SUMMARY:
This is a prospective, observational, monocentric, phase II (exploratory) cohort study aiming to describe the evolutionary profile of the initial volume of glucose distribution (IDVG) during the first four days of management of severely burned patient.

DETAILED DESCRIPTION:
In the early phase, severe burns induce a state of hypovolaemic shock linked to inflammation and a capillary leak syndrome, responsible for the formation of a voluminous third sector. Initial resuscitation of burn patients is based on an assessment of filling requirements using the Parkland formula, which takes into account the patient's weight and the percentage of burned skin surface. This haemodynamic resuscitation oscillates between a risk of underfilling, responsible for hypovolaemia with low cardiac output and leading to excess mortality, and a state of hydric hyperinflation responsible for numerous complications such as respiratory distress, cardiac failure, abdominal compartment syndrome, and even excess mortality. The necessary adaptation of vascular filling rates is usually achieved by monitoring clinical parameters such as diuresis, or biological parameters such as arterial lactate or haematocrit. More advanced haemodynamic monitoring may be applied in addition, but the targets chosen and their numerical objectives remain to be validated. Due to the burn-induced capillary leak syndrome, quantification of extracellular (intra- and extravascular) fluid volume (ECFV) could be a relevant marker of fluid overload status in severely burned patients. ECFV can be estimated using intravenous glucose. Glucose is distributed throughout the extracellular fluid compartment within a few minutes, and defines an initial volume of glucose distribution (IDVG) proportional to the ECFV. This measurement has been validated in healthy individuals and in various pathological conditions. In intensive care patients, the values are between 3.1 and 4.8 L/m2.

To the best of our knowledge, no study has assessed variations in ECV measured by the LVDI in severely burned patients in the early phase of intensive care. Understanding these variations could make a definite contribution to the adaptation of perfused fluid volumes.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Patients hospitalized with burns of at least 30% of body surface area

  * By a thermal mechanism
  * At the CHR Metz-Thionville burn center
  * managed within the 8 hours post-burn
* Patient affiliated to a social security scheme
* Written consent obtained from the patient (or from the trusted person, family or relatives if the patient is unable to sign/express consent) or emergency inclusion if the patient is unable to express consent and neither the trusted support person nor any member of the family or relatives is present at the time of inclusion.

Exclusion Criteria:

* Diabetic patients on insulin
* Patient with a CONTRAINDICATION to GLUCOSE 30% PROAMP, solution for injection
* Patients with pre-hospital cardiac arrest
* extra corporeal circulation patient: Extra Corporeal Membranous Oxygenation (ECMO) or Extra Corporeal Life Support (ECLS) or CRRT (Continuous Renal Replacement Therapy)
* patient without a central venous line or arterial catheter
* Patient moribund or immediately subject to therapeutic limitation
* Impossibility of trans-pulmonary thermodilution monitoring (vascular access difficulties)
* Pregnant, parturient or breast-feeding women
* Patient under guardianship, curatorship or safeguard of justice
* Cognitive impairment or language barrier

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-11-28 (Actual); Primary Completion 2027-03-28 (Estimated); Study Completion 2027-03-28 (Estimated)

PRIMARY OUTCOMES:
Description of the mean values of the initial volume of glucose distribution (IDVG) | on admission, at Hours 4, 8, 16, 24, 48, 72 and 96 post-burn
  The IDVG is calculated according to the method described by Hitota et al. A reference blood glucose level is measured on an arterial blood sample (arterial catheter) by a blood glucose meter. A bolus of 5 g of glucose is injected into a central venous line over 30 seconds.
  A second blood glucose level is measured 3 minutes after the end of the injection.
  The difference between the two blood glucose levels is recorded as d[glu] in mg/dl.
  IDVG = 24.4 x e(-0.0298 * d[glu]) + 2.7 in liters

SECONDARY OUTCOMES:
Study of correlations between initial distribution volume of glucose (IDVG), intra-thoracic blood volume (ITBV) and extra-vascular lung water (EVLW). | on admission, at Hours 4, 8, 16, 24, 48, 72 and 96 post-burn
  ITBV (intra-thoracic blood volume) and EVLW (extra-vascular lung water) measured at the same time as IDVG, using the PiCCO device and trans-lung dilution of a thermal indicator (cold saline).
Study of correlations between IDVG and body surface area (BSA) | at hospital admission
  Body surface area assessed on admission according to Wallace method
Study of correlations between IDVG and water intake and input/output balance | on admission, at Hours 4, 8, 16, 24, 48, 72 and 96 post-burn
  Water intake and input/output balance (water intake minus diuresis)
Study of correlations between IDVG at H24 to H48 and mortality | at Hours 24 and 48 post-burn
  In-hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: Serge LE TACON, MD, Principal Investigator — CHR Metz Thionville Hopital de Mercy
Locations (1):
- CHR Metz-Thionville/Hopital de Mercy, Metz, France

IPD SHARING:
Plan to Share IPD: No